CLINICAL TRIAL: NCT05132816
Title: High Resolution Manometry After Partial Fundoplication for Gastro-oesophageal Reflux: Does the Ineffective Preoperative Oesophageal Motility Change Postoperatively?
Brief Title: High Resolution Manometry After Partial Fundoplication for Gastro-oesophageal Reflux
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Urs Zingg (Other)
Responsible Party: Sponsor-Investigator, Prof Urs Zingg, Prof. Dr., Spital Limmattal Schlieren
Organization: Spital Limmattal Schlieren (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-01536
Record Dates: First submitted 2021-10-14; First posted 2021-11-24 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Gastroesophageal Reflux; Esophageal Motility Disorders; Upper Gastrointestinal Disorder
MeSH Terms: conditions — Gastroesophageal Reflux; Esophageal Motility Disorders; Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main arm (Experimental)
  Interventions: Diagnostic Test: high-resolution manometry

INTERVENTIONS:
Diagnostic Test: high-resolution manometry — High-resolution manometry is an outpatient examination and part of our routine diagnostic or pre-operative evaluation in GERD.
  A thin catheter is placed through the nose into the esophagus, local anaesthesia can be used if the patient experiences a discomfort. Once the tip of the manometry catheter is placed below the esophagogastric junction, the patient is asked to take in water and bread. In rest and during deglutition, pressure measurements are registered with the manometry catheter, allowing the investigator to detect IEM. The examination takes about 1.5 hours. The manometry is a standard and routine intervention being performed for over 30 years with minimal risks.
  The GSRS questionnaire pre- and postoperatively is part of our standard workup, no additional assessment for this study is needed.
  Other Names: Gastrointestinal Symptom Rating Scale (GSRS) - questionnaire

SUMMARY:
This is a combined retro- and prospective, monocentric study. All patients who underwent or are planned for laparoscopic partial fundoplication (180° anterior or 270° posterior) between 2020-2023 are assessed for preoperative ineffective esophageal motility (IEM).

The main hypothesis is, that preoperative oesophageal motility disorders, especially hypo-contractility or failed peristalsis, are caused by gastro-oesophageal reflux. Therefore, postoperative manometry after partial wrap fundoplication (270° posterior, 180° anterior) shows a decrease in comparison to preoperative motility disorders.

The primary objective of this study is to examine the postoperative esophageal motility in patients with known preoperative motility disorders.

Secondary endpoints are the presence of other oesophageal motility disorders pre- vs. postoperatively (including new onset disorders), the assessment of the Gastrointestinal Symptom Rating Scale (GSRS) pre- vs. postoperatively, and more.

If IEM is present preoperatively, patients are contacted at least 1 year after surgery and will be informed about the study and asked to participate. In case of agreement, they are invited to the study site. They undergo high-resolution manometry 18-24 months postoperatively (study intervention).

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Ineffective esophageal motility disorder according the Chicago classification (7), defined as ≥ 7/10 (70%) of swallows with weak contraction (distal contraction interval (DCI) between 100mmHg/s/cm and less than 450 mmHg/s/cm) or ≥ 5/10 (50%) of swallows with failed peristalsis (DCI <100mgHg/s/cm)Performance of partial fundoplication (180° anterior or 270° posterior) at Spital Limmattal
* Informed Consent as documented by signature

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Normal preoperative esophageal motility
* Other specifically defined esophageal motility disorders such as Nutcracker or Jackhammer esophagus
* Preoperative presence of a hiatal hernia with migration of >20% of stomach in the chest
* Revisional surgery (after other procedures for reflux or at the hiatus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of persistent postoperative IEM | 1-2 years postoperatively
  The primary endpoint is the incidence of persistent postoperative ineffective motility according to the Chicago classification, defined as ≥ 7/10 (70%) of swallows with weak contraction (distal contraction interval (DCI) between 100mmHg/s/cm and less than 450 mmHg/s/cm) or ≥ 5/10 (50%) of swallows with failed peristalsis (DCI <100mgHg/s/cm), measured in a high-resolution manometry with multiple swallows in patients having undergone laparoscopic partial-wrap 270° posterior or 180° anterior fundoplication.

SECONDARY OUTCOMES:
Presence of other oesophageal motility disorders | 1-2 years postoperatively
  Presence of other oesophageal motility disorders pre- vs. postoperatively (including new onset disorders) measured in a high-resolution manometry with multiple swallows in patients having undergone laparoscopic partial-wrap 270° posterior or 180° anterior fundoplication.
GSRS | 1-2 years postoperatively
  Gastrointestinal Symptom Rating Scale (GSRS) pre- vs. postoperatively. The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Spital Limmattal, Schlieren, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
The sharing of IPD is not planned.